CLINICAL TRIAL: NCT03842345
Title: Cross-sectional Evaluation of Psychiatric Population With DELPhI- Characterization of Psychiatric Conditions
Brief Title: DELPhI Evaluation of Psychiatric Conditions
Status: Withdrawn | Type: Observational
Why Stopped: Study was withdrawn due to recruitment difficulties
Sponsor: QuantalX Neuroscience (Industry)
Responsible Party: Sponsor
Other Study IDs: 605
Record Dates: First submitted 2019-02-06; First posted 2019-02-15 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2019-02

CONDITIONS: Major Depressive Disorder; Bi-Polar Disorder; ADHD; Schizophrenia; OCD; Ptsd; Healthy
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Attention Deficit Disorder with Hyperactivity; Schizophrenia; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Psychiatric patients: Major depression, Bi-polar, schizophrenia, ADHD, OCD, PTSD
- healthy controls: young healthy controls to serve as norm.

SUMMARY:
DELPhI acquisition and analysis software, a QuantalX Neuroscience development, which is designed to measure, analyze, and display brain electrical activity of human electroencephalogram (EEG), to transcranial magnetic stimulation (TMS), will be used to evaluate different psychiatric conditions.

DETAILED DESCRIPTION:
Psychiatric conditions requiring pharmaceutical treatment include Schizophrenia and other psychotic disorders, Major depressive disorder, Bi-polar disorder, Post Traumatic Stress Disorder, Obsessive Compulsive Disorder and anxiety disorders. To date none of the psychiatric conditions mentioned diagnosis' relies on an imaging or other quantitative technique. Diagnosis and treatment prescription in the psychiatric clinic still relies on subjective reports and physician assessment of symptoms. Trans-cranial magnetic stimulation (TMS) is a noninvasive brain stimulation method that allows to study human cortical function In-vivo. Using TMS for examining human cortical functionality is enhanced by combining TMS with simultaneous registration of electroencephalograph (EEG). EEG provides an opportunity to directly measure the cerebral response to TMS, measuring the cortical TMS Evoked potential (TEP), is used to assess cerebral reactivity across wide areas of neo-cortex. Studies integrating TMS with EEG (TMS-EEG) have shown that TMS produces waves of activity that reverberate throughout the cortex. and that are reproducible and reliable thus providing direct information about cortical excitability and connectivity with excellent time resolution. By evaluating the propagation of evoked activity in different behavioral states and in different tasks, TMS-EEG has been used to causally probe the dynamic effective connectivity of human brain networks.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female patients between the age of 18-80 years old.
2. Patients willing to participate with all of the study procedures and sign informed consent form.
3. A clinical diagnosis of psychiatric condition that requires medication or other intervention (such as brain stimulation or psychological treatment).-study groups.
4. Without any psychiatric medications or with stable treatment regimen for the last 2 months-study groups..

4.5. A normal neurological exam- control group.

Exclusion criteria:

1. Prior known epileptic episode. 2. History of any neurodegenerative disease. 3. Patients with history of other known brain disorder/pathology. 4. Contraindication to MR imaging.

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: study group: patients diagnosed with either Major depression, Bi-polar disorder, OCD, PTSD, ADHD or Schizophrenia,.without any psychiatric medications or with stable treatment regimen for the last 2 months.
  Control group:
  Eligible consecutive healthy individuals, recruited through advertisements spread in campuses and clinics.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
comparison of DELPhI parameter of Plasticity in psychiatric population to healthy norms. | through study completion, an average of 1 year
  Comparison of DELPhI parameters of Plasticity in patients, in comparison to healthy norms. Parameters will be analyzed for their temporal and special components.
comparison of DELPhI parameter of Connectivity in psychiatric population to healthy norms. | through study completion, an average of 1 year
  Comparison of DELPhI parameters of Connectivity in patients, in comparison to healthy norms. Parameters will be analyzed for their temporal and special components.

SECONDARY OUTCOMES:
correlation between DELPhI parameters and symptom severity. | through study completion, an average of 1 year
  Self-control analysis of the change in DELPhI parameters following change in treatment prescription or any other treatment at different time points compared to base-line. Correlation to symptom severity will be assessed.
Cluster analysis of Plasticity and connectivity in relation to medical treatment and clinical diagnosis. | through study completion, an average of 1 year.
  Cluster subjects by each plasticity and connectivity vs. medical treatment and clinical diagnosis.
characterization of the change in Plasticity following change of treatment regimen | through study completion, an average of 1 year.
  characterization of the change in Plasticity of Plasticity following change of treatment regimen.
characterization of the change in Connectivity following change of treatment regimen | through study completion, an average of 1 year.
  characterization of the change in Connectivity following change of treatment regimen.

IPD SHARING:
Plan to Share IPD: No